CLINICAL TRIAL: NCT01881763
Title: Comparing Therapeutic Efficacy and Cognitive Side Effects of Electroconvulsive Therapy (ECT) Using Ketamine Versus Methohexital Anesthesia
Brief Title: Ketamine as an Augmentation Strategy for Electroconvulsive Therapy (ECT) in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-127
Record Dates: First submitted 2013-05-07; First posted 2013-06-20 (Estimated); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Unipolar Depression; Bipolar Depression
Keywords: Electroconvulsive Therapy; Ketamine; anesthesia; depression; unipolar; bipolar
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Depression | interventions — Ketamine; Methohexital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Participants will be randomized 1:1 to either Ketamine (experimental condition) or Methohexital anesthesia (active comparator)
  Interventions: Drug: Ketamine
- Methohexital (Active Comparator): Participants will be randomized 1:1 to either Ketamine (experimental condition) or Methohexital anesthesia (active comparator)
  Interventions: Drug: Methohexital

INTERVENTIONS:
Drug: Ketamine — Ketamine 1-2 mgr/ kg IV
  Other Names: Ketalar
  Arms: Ketamine
Drug: Methohexital — Methohexital 0.5-1mg/kg IV
  Other Names: Brevatol
  Arms: Methohexital

SUMMARY:
The study aims to compare outcomes of Electroconvulsive Therapy (ECT) using ketamine versus methohexital anesthesia in depressed patients. The investigators hypothesize that patients who receive ketamine anesthesia during ECT will achieve remission status faster than those receiving methohexital anesthesia. Also, at the end of the ECT course subjects will display fewer cognitive side effects compared to those treated with methohexital anesthesia.

DETAILED DESCRIPTION:
Despite major advances in the treatment of mood disorders, depression remains a serious public health problem. Delayed onset of response and lack of efficacy in a significant portion of patients are the limitations of pharmacotherapy. Electroconvulsive therapy (ECT) has been shown to provide fast amelioration of depressive symptoms and its efficacy is reported to be 65 to 85%. However, one of the main limiting factors for its use is the cognitive impairment, which is directly related to the number of ECT sessions.

There is increased evidence for the mediation of glutamate in the pathophysiology of depression, as suggested by the potential antidepressant effect of drugs that modulate glutamate transmission. Open studies and recent case reports demonstrate a rapid antidepressant effect of intravenous ketamine - a non-competitive antagonist at the glutamate N-methyl-D-aspartate (NMDA) receptor. Ketamine is a general anesthetic used commonly for procedural sedation. Ketamine has no anticonvulsant properties. It is used as an alternative to methohexital - a barbiturate with anticonvulsant properties - in patients with high seizure threshold. A recent open non-randomized trial by Okamoto shows a faster response when ECT is given with ketamine anesthesia. In a recent review Gregory-Roberts et al suggest that available evidence in animals and humans supports the prediction that ketamine could effectively prevent ECT -induced persistent retrograde amnesia and improve or hasten therapeutic response.

We propose a double-blind randomized controlled pilot study to measure both therapeutic efficacy and cognitive side effects of ECT using ketamine compared to methohexital - the gold standard anesthetic in ECT - in depressed patients.

Thirty patients who are scheduled to receive an acute course of ECT for major depressive episode. Inpatients and outpatients will be screened by the ECT psychiatrists who participate in this study. Patients who are able and willing to provide written informed consent will be randomly assigned on a 1:1 ratio to receive either a course of bifrontal ECT using ketamine 1-2 mg/kg or methohexital anesthesia0.5-1.0 mg/kg. Subjects will receive a standard acute course of ECT (3X/week. Raters and subjects will be masked to group assignment.

Parallel with these procedures we will also collect magnetic resonance imaging (MRI) data on these subjects. The timeline of neuroimaging and it relation to ECT is a baseline MRI prior to first ECT, and then a follow up MRI after the first ECT (< 36hrs after), and a final MRI after 9 ECTs or if patient remits. All subjects will receive structural (i.e. diffusion tensor imaging and spectroscopy) and functional MRI exams.

In addition to the imaging procedures detailed above, we also plan to acquire imaging data on healthy individuals with similar timeline. Healthy volunteers will be scanned three times; the first and second scans will be 24-48 hours apart, while the second and third scans will be two weeks apart. The imaging sessions will follow the same protocol as in the patients. The collection of control data is necessary in order to demonstrate that imaging findings are not due to acclimatization to scanner environment or other confounding sources. Compensation for participating in the MRI component is $75 per MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 70 years of age
2. Diagnostic Statistical Manual (DSM) IV diagnosis of Major Depression (296.3), unipolar without psychotic features or Bipolar I or Bipolar II Depression without psychotic features confirmed by Structured Clinical Interview for DSM-IV (SCID-IV) interview
3. Pretreatment 24-item Hamilton Rating Scale for Depression score > 21
4. Subjects must have an initial score of at least 20 on the Montgomery-Asbergers Depression Rating Scale (MADRS) at screen
5. ECT is clinically indicated
6. Patient is competent to provide informed consent

Exclusion Criteria:

1. Lifetime DSM-IV diagnosis of schizophrenia, schizoaffective disorder, psychotic depression or any other psychotic disorder as defined in the DSM-IV
2. Current (within the last year) diagnosis of anxiety disorder, obsessive- compulsive disorder, or eating disorder that precedes the onset of the current episode of depression
3. Current diagnosis of delirium, dementia, or amnestic amnesiac disorder
4. Diagnosis of Mental Retardation
5. Baseline Mini Mental State Exam (MMSE) score < 21 or a total score falling two standard deviations below the age- and education-adjusted mean, whichever is less
6. Any active general medical condition or central nervous system (CNS) disease which can affect cognition or response to treatment
7. Current (within the past three months) diagnosis of active substance dependence, or active substance abuse within the past week
8. Lifetime history of ketamine or phencyclidine (PCP) abuse or dependence
9. ECT within three months
10. The presence of any known or suspected contraindication to methohexital or ketamine including but not limited to known allergic reactions to these agents, uncontrolled hypertension, arrhythmia, severe coronary artery disease and porphyria
11. Pregnancy
12. Status 4 or greater according to the criteria of the American Society of Anesthesiologists
13. MRI contraindications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Petrides, M.D., Principal Investigator — The Zucker Hillside Hospital
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kellner CH, Knapp RG, Petrides G, Rummans TA, Husain MM, Rasmussen K, Mueller M, Bernstein HJ, O'Connor K, Smith G, Biggs M, Bailine SH, Malur C, Yim E, McClintock S, Sampson S, Fink M. Continuation electroconvulsive therapy vs pharmacotherapy for relapse prevention in major depression: a multisite study from the Consortium for Research in Electroconvulsive Therapy (CORE). Arch Gen Psychiatry. 2006 Dec;63(12):1337-44. doi: 10.1001/archpsyc.63.12.1337. PMID 17146008
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Okamoto N, Nakai T, Sakamoto K, Nagafusa Y, Higuchi T, Nishikawa T. Rapid antidepressant effect of ketamine anesthesia during electroconvulsive therapy of treatment-resistant depression: comparing ketamine and propofol anesthesia. J ECT. 2010 Sep;26(3):223-7. doi: 10.1097/YCT.0b013e3181c3b0aa. PMID 19935085
- [Background] Gregory-Roberts EM, Naismith SL, Cullen KM, Hickie IB. Electroconvulsive therapy-induced persistent retrograde amnesia: could it be minimised by ketamine or other pharmacological approaches? J Affect Disord. 2010 Oct;126(1-2):39-45. doi: 10.1016/j.jad.2009.11.018. Epub 2010 Jan 8. PMID 20060172
- [Background] Sanacora G, Rothman DL, Mason G, Krystal JH. Clinical studies implementing glutamate neurotransmission in mood disorders. Ann N Y Acad Sci. 2003 Nov;1003:292-308. doi: 10.1196/annals.1300.018. PMID 14684453
- [Background] Ostroff R, Gonzales M, Sanacora G. Antidepressant effect of ketamine during ECT. Am J Psychiatry. 2005 Jul;162(7):1385-6. doi: 10.1176/appi.ajp.162.7.1385. No abstract available. PMID 15994728
- [Derived] Dean RL, Marquardt T, Hurducas C, Spyridi S, Barnes A, Smith R, Cowen PJ, McShane R, Hawton K, Malhi GS, Geddes J, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with bipolar disorder. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD011611. doi: 10.1002/14651858.CD011611.pub3. PMID 34623633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine | Methohexital
Started | 16 | 15
Completed | 10 | 11
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Methohexital | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.01 (15.04) | 48.34 (9.27) | 48.17 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HRSD) Improvement
Description: The items mostly range from a score of 0-4 but there are some questions that range from a score of 0-2. The maximum total score that can be reported is 76 and the lowest score is 0. Higher values represent a worse outcome. Items are summed together to compute the total score. Remission is defined as two consecutive Hamilton Rating Scale for Depression, 24 items (HRSD-24) scores < 10, and HRSD-24 total score does not increase > 3 points on the second consecutive HRSD-24, or remains < 6 at the last two consecutive treatments. HRSD-24 scores are used to define remission.
Time Frame: Days required to achieve remission (on average 3-4 weeks)
Measure: Mean (Standard Deviation); unit: HRSD units
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 10 | 11
HRSD units | 7.82 (3.43) | 8.60 (3.72)

2. Secondary Outcome: Cognitive Side Effects of ECT
Description: To determine the cognitive side effects we will use the following neuropsychological battery:
  * Mini- Mental State Examination (MMSE),
  * Postictal Recovery of Orientation,
  * Rey Auditory Verbal Learning Test (RAVLT)
  * Autobiographical Memory Interview - Short Form (AMI - SF),
  * Subjective Memory Questionnaire (SMQ),
  * Reading subtest of the Wide Range Achievement Test, 3rd Edition (WRAT-3),
  * The Stroop Color Word Test (SCWT) (Golden version),
  * Trail Making Test Part A & B,
  * Wechsler Adult Intelligence Test-Third Edition (WAIS-III), Digit Span Subtest,
  * WAIS-III Digit Symbol,
  * Controlled Oral Word Association Test (COWAT),
  * N-Back test
Time Frame: Neuropsychological Battery: Changes from baseline to the end of the ECT course (on average 3-4 weeks)
Population: Data was not collected and the outcome cannot be reported. A total of 0 participants were analyzed due to slower than anticipated recruitment for this study therefore, we were not able to recruit a sufficient number of subjects for statistical analysis prior to the end of the funding period.
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Resting Stated Functional Magnetic Resonance Imaging (rs fMRI)
Description: To use resting state and task related fMRI to identify ECT related functional network changes in the brain. Using resting state fMRI before and after ECT, we will (a) identify networks modulated by ECT (defined as a decrease or increase in functional connectivity from baseline to follow up scans), and we will (b) follow up their expression in the upcoming weeks, we will (c) identify functional networks of the brain which are correlated with superior clinical ECT outcome and we will (d) identify functional networks of the brain which are correlated with side effect profiles.
Time Frame: Changes from baseline to the end of ECT course (approximately 3-4 weeks)
Population: as for outcome 2
Arm/Group | Ketamine | Methohexital
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The study duration was variable depending upon subject response, but no more than 15 ECT treatments over approximately 5 weeks occurred.
Arm/Group | Ketamine | Methohexital
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT01881763/Prot_SAP_000.pdf